CLINICAL TRIAL: NCT00396266
Title: Treatment With AMD3100 in Non-Hodgkin's Lymphoma and Multiple Myeloma Patients to Increase the Number of Peripheral Blood Stem Cells When Given a Mobilizing Regimen of G-CSF
Brief Title: AMD3100 (Plerixafor) Given to NHL and MM Patients to Increase the Number of PBSCs When Given a Mobilizing Regimen of G-CSF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMD3100-C201
Record Dates: First submitted 2006-11-02; First posted 2006-11-06 (Estimated); Results first posted 2010-11-25 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-02

CONDITIONS: Multiple Myeloma; Lymphoma, Non-Hodgkin
Keywords: Non-Hodgkin's Lymphoma; Multiple Myeloma; stem cell mobilization; AMD3100; autologous transplantation
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, Non-Hodgkin | interventions — Granulocyte Colony-Stimulating Factor; plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-Hodgkin's Lymphoma (NHL) (Experimental): Participants with NHL were mobilized with granulocyte colony-stimulating factor (G-CSF) 10 µg/kg/day for 4 days. Plerixafor 240 µg/kg was given the evening of day 4 and G-CSF given the next morning followed by apheresis. Evening doses of plerixafor and morning doses of G-CSF followed by apheresis continued for up to a maximum of 5 aphereses or until ≥ 5*10^6 CD34+ cells/kg were collected.
  Interventions: Drug: G-CSF Plus Plerixafor
- Multiple Myeloma (MM) (Experimental): Participants with MM were mobilized with granulocyte colony-stimulating factor (G-CSF) 10 µg/kg/day for 4 days. Plerixafor 240 µg/kg was given the evening of day 4 and G-CSF given the next morning followed by apheresis. Evening doses of plerixafor and morning doses of G-CSF followed by apheresis continued for up to a maximum of 5 aphereses or until ≥ 5*10^6 CD34+ cells/kg were collected.
  Interventions: Drug: G-CSF Plus Plerixafor

INTERVENTIONS:
Drug: G-CSF Plus Plerixafor — Participants underwent mobilization with G-CSF 10 µg/kg/day for 4 days, administered by subcutaneous injection (SC) injection each morning. On the evening of Day 4, participants received a dose of plerixafor 240 µg/kg, administered by SC injection. On Day 5, participants returned to the clinic and received a morning dose of G-CSF 10 µg/kg and underwent apheresis approximately 10 to 11 hours after the dose of plerixafor (within 60 minutes after administration of G-CSF). Participants continued to receive an evening dose of plerixafor followed the next day by a morning dose of G-CSF and apheresis for up to a maximum of 5 aphereses or until ≥ 5*10^6 CD34+ cells/kg were collected.
  Other Names: Mozobil; AMD3100

SUMMARY:
This study evaluates the safety and efficacy of plerixafor given in addition to granulocyte-colony stimulating factor (G-CSF) for collection of peripheral blood stem cells (PBSCs) for autologous transplantation in patients with non-Hodgkin's lymphoma (NHL) and multiple myeloma (MM). Efficacy outcomes include evaluation of fold increase in circulating CD34+ cells from just before the first plerixafor injection to 10-11 hours post plerixafor (just before apheresis) and assessment of successful polymorphonuclear leukocyte (PMN) engraftment after transplantation. Data from this protocol will assist in the determination of the dosing schedule for future studies.

DETAILED DESCRIPTION:
Participants with NHL and MM who have undergone prior cyto-reductive chemotherapy, are to be autologously transplanted, and meet the inclusion/exclusion criteria are eligible to enter the study. The only change to the standard of care is the addition of plerixafor to a granulocyte colony-stimulating factor (G-CSF) mobilization regimen on the day prior to apheresis. Participants will undergo mobilization with G-CSF (10 mcg/kg each day) and will receive plerixafor (240 mcg/kg) in the evening prior to apheresis. Participants will undergo apheresis for up to 5 consecutive days in order to collect the target number of CD34+ stem cells (≥ 5*10^6 CD34+ cells/kg for either single or tandem transplant). After apheresis, all participants will be treated with high-dose chemotherapy in preparation for transplantation. Participants will be transplanted with cells obtained from the G-CSF and plerixafor mobilization regimen. The increase in CD34+ cells in the peripheral blood from the time of the plerixafor dose to just prior to apheresis and the number of CD34+ cells in the apheresis product will be measured. Success of the transplantation(s) will be evaluated by the time to engraftment of polymorphonuclear leukocytes (PMN). A subpopulation will have pharmacokinetic and pharmacodynamic analysis done.

This study was previously posted by AnorMED, Inc. In November 2006, AnorMED, Inc. was acquired by Genzyme Corporation. Genzyme Corporation is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-Hodgkin's lymphoma (NHL) or multiple myoloma (MM) eligible for autologous transplantation
* No more than 3 prior regimens of chemotherapy
* More than 4 weeks since last cycle of chemotherapy. Patient recovered from all acute toxic effects of prior chemotherapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* White blood cell (WBC) count >3.0*10^9/L
* Absolute polymorphonuclear cells (PMN) count >1.5*10^9/L
* Platelet (PLT) count >100*10^9/L
* Serum creatinine <=2.2 mg/dL
* Serum glutamic oxaloacetic transaminase (SGOT), serum glutamic pyruvic transaminase (SGPT) and total bilirubin <2 x upper limit of normal (ULN)
* Left ventricle ejection fraction >45% by normal echocardiogram or multiple-gated acquisition (MUGA) scan
* Forced expiratory volume of the lung in the first second (FEV1) >60% of predicted or diffusing capacity of the lung for carbon monoxide (DLCO) >45% of predicted
* Negative for human immunodeficiency virus (HIV) type 1
* Women of child bearing potential agreed to use an approved form of contraception.

Exclusion Criteria:

* • Patients who have failed previous collections

  * Brain metastases or carcinomatous meningitis
  * History of ventricular arrhythmias
  * A co-morbid condition which, in the view of the investigator, renders the patient at high risk for treatment complications
  * A residual acute medical condition resulting from prior chemotherapy
  * Acute infection
  * Fever (temp >38°C/100.4°F)
  * Patients whose actual body weight exceeds 150% of their ideal body weight
  * History of paresthesias (at least Grade 2)
  * Patients who previously received experimental therapy within 4 weeks of enrolling in this study or who are currently enrolled in another experimental study during the mobilization period
  * Positive pregnancy test in female patients
  * Lactating females
  * Patients of child-bearing potential unwilling to implement adequate birth control.
  * Patients who have deterioration of their clinical status or laboratory parameters between the time of enrolment and transplant (such that they no longer meet entry criteria) may be removed from study at the discretion of the treating physician, principal investigator, or sponsor.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2005-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Genzyme, a Sanofi Company
Locations (2):
- Canada (2):
  - Tom Baker Cancer Center, Calgary, Alberta
  - Vancouver General Hospital, BC Cancer Agency, Vancouver, British Columbia

REFERENCES:
- [Result] Stewart DA, Smith C, MacFarland R, Calandra G. Pharmacokinetics and pharmacodynamics of plerixafor in patients with non-Hodgkin lymphoma and multiple myeloma. Biol Blood Marrow Transplant. 2009 Jan;15(1):39-46. doi: 10.1016/j.bbmt.2008.10.018. PMID 19135941

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Non-Hodgkin's Lymphoma (NHL) | Multiple Myeloma (MM)
Started | 8 | 14
Completed | 8 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-Hodgkin's Lymphoma (NHL) | Multiple Myeloma (MM) | Total
Number analyzed (Participants) | 8 | 14 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (8.7) | 57.5 (10.3) | 57.6 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 5 | 10 | 15

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants Who Had a ≥ 2-fold Increase in Circulating CD34+ Cells
Description: To determine if NHL and MM patients mobilized with G-CSF (10 µg/kg QD) plus plerixafor will have a ≥2-fold increase in circulating CD34+ cells from time 0 to 11 hours after a dose of plerixafor.
Time Frame: Time 0 to 11 hours after the first dose of plerixafor
Population: The intent-to-treat population (defined as participants who received at least 1 dose of plerixafor).
  One participant excluded from the analysis because data was missing.
Measure: Number; unit: participants
Groups:
- Total: All patients.
Arm/Group | Non-Hodgkin's Lymphoma (NHL) | Multiple Myeloma (MM) | Total
Number analyzed (Participants) | 8 | 13 | 21
participants
  ≥ 2-fold Increase | 8 | 13 | 21
  < 2-fold Increase | 0 | 0 | 0

2. Secondary Outcome: Number of Transplants Resulting In Polymorphonuclear Leukocyte (PMN) Engraftment by Day 12 But No Later Than Day 21 Post-Transplant
Description: Participants were monitored for polymorphonuclear leukocyte (PMN) engraftment as per the local standard of care. The target for engraftment was 12 days after PBSC transplant and no transplant taking longer than 21 days for engraftment.
Time Frame: 2 months
Population: Intent to treat population of participants who had transplants. One participant received a tandem transplant.
Measure: Number; unit: number of transplants
Units Other Than Participants: transplants
Arm/Group | Non-Hodgkin's Lymphoma (NHL) | Multiple Myeloma (MM) | Total
Number analyzed (Participants) | 8 | 14 | 22
Number analyzed (transplants) | 8 | 15 | 23
number of transplants
  ≤ Day 12 | 7 (1.5) | 10 (2.8) | 17
  Day 13 to Day 21 | 1 | 5 | 6
  ≥ Day 22 | 0 | 0 | 0

3. Secondary Outcome: Tumor Cell Mobilization in Non-Hodgkin's Lymphoma (NHL) Participants Following Plerixafor Treatment
Description: In a subpopulation of NHL participants, the mobilization of NHL cells was to be evaluated. None of the samples were analyzed due to sample degradation.
Time Frame: Prior to the first (Day 4) and last dose of plerixafor, immediately prior to each apheresis, and 24 hours after the last apheresis.
Population: This analysis was not performed due to sample degradation.
Arm/Group | Non-hodgkin's Lymphoma (NHL)
Number analyzed (Participants) | 0

4. Secondary Outcome: Single-dose Maximum Observed Concentration of Plerixafor (Cmax)
Description: Evaluation of Cmax following a single dose of 240 µg/kg plerixafor administered after 4 days of G-CSF mobilization. Cmax was determined from direct observation of the data.
Time Frame: Day 5 - 0 to 10 hours post-first plerixafor dose.
Population: Pharmacokinetic analysis was performed on a subgroup of participants from both treatment arms (5 NHL and 8 MM).
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- PK Subgroup: Subgroup of 13 participants (5 NHL and 8 MM) for which a pharmacokinetic (PK) profile was analyzed. Participants were mobilized with granulocyte colony-stimulating factor (G-CSF) 10 µg/kg/day for 4 days, followed by plerixafor 240 µg/kg the evening of day 4.
Arm/Group | PK Subgroup
Number analyzed (Participants) | 13
ng/mL | 926 (237)

5. Secondary Outcome: Single-dose Time to Maximum Concentration of Plerixafor (Tmax)
Description: Evaluation of Tmax following a single dose of 240 µg/kg plerixafor administered after 4 days of G-CSF mobilization. Tmax was determined from direct observation of the data.
Time Frame: Day 5 - 0 to 10 hours post-first plerixafor dose
Population: Pharmacokinetic analysis was performed on a subgroup of participants from both treatment arms (5 NHL and 8 MM).
Measure: Median (Full Range); unit: hours
Arm/Group | PK Subgroup
Number analyzed (Participants) | 13
hours | 0.5 (0.2) [0.3 to 1.0]

6. Secondary Outcome: Single-dose Half-life of Plerixafor (T1/2)
Description: Evaluation of T1/2 following a single dose of 240 µg/kg plerixafor administered after 4 days of G-CSF mobilization. T1/2 was determined from non-compartmental analysis.
Time Frame: Day 5 - 0 to 10 hours post-first plerixafor dose.
Population: Pharmacokinetic analysis was performed on a subgroup of participants from both treatment arms (5 NHL and 8 MM).
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PK Subgroup
Number analyzed (Participants) | 13
hours | 5.1 (2.2)

7. Secondary Outcome: Single-dose Area Under the Concentration-time Curve of Plerixafor From Time 0 to 10 Hours Post-dose (AUC0-10)
Description: Evaluation of AUC0-10 following a single dose of 240 µg/kg plerixafor administered after 4 days of G-CSF mobilization. AUC0-10 was determined from non-compartmental analysis.
Time Frame: Day 5 - 0 to 10 hours post-first plerixafor dose.
Population: Pharmacokinetic analysis was performed on a subgroup of participants from both treatment arms (5 NHL and 8 MM).
Measure: Mean (Standard Deviation); unit: ng•h/mL
Arm/Group | PK Subgroup
Number analyzed (Participants) | 13
ng•h/mL | 3594 (697)

8. Secondary Outcome: Single-dose Apparent Clearance of Plerixafor (CL/F)
Description: Evaluation of Cl/F following a single dose of 240 µg/kg plerixafor administered after 4 days of G-CSF mobilization. Cl/F was determined from non-compartmental analysis.
Time Frame: Day 5 - 0 to 10 hours post-first plerixafor dose.
Population: Pharmacokinetic analysis was performed on a subgroup of participants from both treatment arms (5 NHL and 8 MM).
Measure: Mean (Standard Deviation); unit: mL/hour
Arm/Group | PK Subgroup
Number analyzed (Participants) | 13
mL/hour | 4767 (1063)

9. Primary Outcome: Number of Participants in Overall Safety Summary of Treatment Emergent Adverse Events (TEAE)
Description: Number of participants with treatment emergent adverse events (TEAEs) collected from Day 1 (start of G-CSF mobilization) to the day before starting chemotherapy. AEs were graded by the investigator using the World Health Organization (WHO) Adverse Event Grading Scale and were assessed for severity (mild, moderate, severe) and relatedness to study treatment (5 point scale from 'not related' to 'definitely related').
Time Frame: Day 1 to approximately Day 38 (before start of chemotherapy)
Population: Safety population - all participants who received at least 1 dose of plerixafor.
Measure: Number; unit: participants
Arm/Group | Non-Hodgkin's Lymphoma (NHL) | Multiple Myeloma (MM) | Total
Number analyzed (Participants) | 8 | 14 | 22
participants
  AE Severity (Mild) | 4 | 8 | 12
  AE Severity (Moderate) | 4 | 6 | 10
  AE Severity (Severe) | 0 | 0 | 0
  AE Relationship to Drug (Not related) | 0 | 0 | 0
  AE Relationship to Drug (Probably not related) | 2 | 3 | 5
  AE Relationship to Drug (Possibly related) | 0 | 5 | 5
  AE Relationship to Drug(Probably related) | 4 | 5 | 9
  AE Relationship to Drug (Definitely related) | 2 | 1 | 3

10. Secondary Outcome: Single-dose Apparent Volume of Distribution of Plerixafor (Vz/F) in NHL and MM Patients
Description: Evaluation of Vz/F following a single dose of 240 µg/kg plerixafor administered after 4 days of G-CSF mobilization. Vz/F was determined from non-compartmental analysis.
Time Frame: Day 5 - 0 to 10 hours post-first plerixafor dose.
Population: Pharmacokinetic analysis was performed on a subgroup of participants from both treatment arms (5 NHL and 8 MM).
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | PK Subgroup
Number analyzed (Participants) | 13
mL | 33668 (10531)

11. Secondary Outcome: Maximum Fold Increase in Peripheral Blood CD34+ Cells From Baseline Following Initial Administration of Plerixafor
Description: A pharmacodynamic evaluation to determine the maximum fold increase in peripheral blood CD34+ cells following the initial administration of plerixafor by measuring the fold increase at time points up to 10 hours post plerixafor relative to baseline (immediately prior to plerixafor).
Time Frame: Day 4 (10 hours post first plerixafor dose)
Population: Pharmacodynamic analysis was performed on a subgroup of participants from both treatment arms (1 NHL and 3 MM). The maximum fold increase was observed at 10 hours for all participants.
Measure: Median (Full Range); unit: ratio
Groups:
- PD Subgroup: Subgroup of 4 patients (3 MM and 1 NHL) for which a pharmacodynamic (PD) profile was analyzed. Participants were mobilized with granulocyte colony-stimulating factor (G-CSF) 10 µg/kg/day for 4 days, followed by plerixafor 240 µg/kg the evening of day 4.
Arm/Group | PD Subgroup
Number analyzed (Participants) | 4
ratio | 4.2 [3.0 to 5.5]

ADVERSE EVENTS:
Time Frame: Treatment emergent AEs covering Day 1 (start of G-CSF Mobilization to the day before starting chemotherapy (approximately Day 38).
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables.
  Each AE table includes events, regardless of reported relationship to study treatment or grade.
Arm/Group | Non-Hodgkin's Lymphoma (NHL) | Multiple Myeloma (MM)
Serious Adverse Events (participants affected / at risk) | 1/8 | 2/14
Other Adverse Events (participants affected / at risk) | 8/8 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-Hodgkin's Lymphoma (NHL) (N=8) | Multiple Myeloma (MM) (N=14)
Catheter site haemorrhage (General disorders) | 1 | 1
Catheter site pain (General disorders) | 0 | 1
Catheter bacteraemia (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-Hodgkin's Lymphoma (NHL) (N=8) | Multiple Myeloma (MM) (N=14)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 7
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 4
Retching (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Catheter site erythema (General disorders) | 1 | 6
Catheter site haematoma (General disorders) | 1 | 0
Catheter site haemorrhage (General disorders) | 0 | 1
Catheter site pain (General disorders) | 2 | 3
Catheter site pruritus (General disorders) | 0 | 1
Catheter site rash (General disorders) | 0 | 1
Catheter site related reaction (General disorders) | 1 | 0
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Chills (General disorders) | 0 | 1
Fatigue (General disorders) | 3 | 6
Influenza like illness (General disorders) | 0 | 1
Injection site bruising (General disorders) | 0 | 1
Injection site erythema (General disorders) | 4 | 6
Injection site irritation (General disorders) | 1 | 1
Injection site pain (General disorders) | 1 | 3
Injection site pruritus (General disorders) | 1 | 2
Injection site swelling (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 3
Swelling (General disorders) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Blood glucose increased (Investigations) | 0 | 1
Heart rate increased (Investigations) | 1 | 0
Urine output increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 6
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 2
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Dizziness (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 3 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 4 | 1
Sensory loss (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 1 | 2
Pallor (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In multi-site studies, PI can publish after Genzyme publishes or 18 months after study completion. PI gives Genzyme a draft 60 days before publication. Genzyme can ask that confidential information be removed, and can defer publication another 60 days upon notifying PI that it will file a patent application on inventions contained in the draft.